CLINICAL TRIAL: NCT04125836
Title: A Phase 3, Open-label, Single-arm, Multi-center Trial to Assess the Long-term Safety of Octreotide Subcutaneous Depot (CAM2029) in Patients With Acromegaly
Brief Title: A Trial to Assess the Long-term Safety of Octreotide Subcutaneous Depot in Patients With Acromegaly
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Camurus AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-19-647; 2019-002190-66 (EudraCT Number)
Record Dates: First submitted 2019-10-11; First posted 2019-10-14 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Acromegaly
Keywords: Acromegaly; octreotide; CAM2029; phase 3
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CAM2029 (octreotide subcutaneous depot) (Experimental): CAM2029 (octreotide subcutaneous depot) 20mg/1.0 mL for 20 mg dose, subcutaneous injection once monthly, 12 months treatment with an option of extension. If down-titration is required, 10mg/0.5 mL for 10 mg dose is available.
  Interventions: Drug: CAM2029 (octreotide subcutaneous depot)

INTERVENTIONS:
Drug: CAM2029 (octreotide subcutaneous depot) — Octreotide subcutaneous depot for monthly injections in acromegaly patients
  Other Names: CAM2029

SUMMARY:
The purpose of this trial is to assess the long-term safety and efficacy of CAM2029 in patients with acromegaly. Patients will be administered CAM2029 subcutaneously once monthly during 12 months. Patients fulfilling trial NCT04076462 will be offered to continue with open-label treatment week 24-52 in this trial. Patients completing the main part of the trial will be offered 52 weeks continued open-label treatment in an extension part.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, ≥18 years at screening
* Able to provide written informed consent to participate in the trial
* Diagnosis of acromegaly by historical evidence of (persistent or recurrent) acromegaly
* Treatment with a stable dose of octreotide LAR or lanreotide ATG for at least 3 months as monotherapy prior to screening
* IGF-1 levels ˃1xULN and ≤2.0xULN at screening or IGF-1 levels ≤1xULN at screening with or without prior pituitary radiotherapy
* Adequate liver, pancreatic, renal and bone marrow functions
* Normal ECG

Exclusion Criteria:

For Roll-over Patients from NCT04076462:

* Unresolved, drug-related serious adverse event (SAE) from the preceding trial
* Patients with a clinically significant or unstable medical or surgical condition that may preclude safe and complete trial participation

For New Patients:

* Have received medical treatment for acromegaly with pasireotide (within 6 months prior to screening), pegvisomant (within 3 months prior to screening), dopamine agonists (within 3 months prior to screening) or other investigational agents (within 30 days or 5 half-lives prior to screening [whichever is longer]
* Patients who usually take octreotide LAR or lanreotide ATG less frequently than every 4 weeks (e.g. every 6 weeks or 8 weeks)
* Patients with compression of the optic chiasm causing any visual field defect for whom surgical intervention is indicated
* Patients who have undergone major surgery/surgical therapy for any cause within 1 month from screening
* Patients who have undergone pituitary surgery within 6 months prior to screening
* Patients who have received prior pituitary irradiation within 3 years prior to screening
* Patients with poorly controlled diabetes mellitus (hemoglobin A1c >8.0%)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2025-04-24 (Actual); Study Completion 2025-04-24 (Actual)

PRIMARY OUTCOMES:
Characterization of adverse events (AEs) | Week 0-52

SECONDARY OUTCOMES:
Proportion of patients with mean IGF-1 levels ≤1xULN and <1.3xULN | Week 50 to 52
Proportion of patients with mean GH levels <2.5 µg/L and <5.0 µg/L | Week 50 to 52
Proportion of patients/partners declared competent by a healthcare professional to administer intervention | Week 0-52
  During patients/partners first three attempts during the trial period of 52 weeks whenever these visits take place
Octreotide plasma concentrations over time | Week 0-52

CONTACTS AND LOCATIONS:
Overall Officials: Diego Ferone, M.D, Principal Investigator — University of Genova Endocrinology Unit
Locations (68):
- United States (12):
  - UCLA Department of Medicine Division of Endocrinology, Los Angeles, California
  - Stanford University Medical Center, Palo Alto, California
  - Prufen Clinical Research LLC, Miami, Florida
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University in St. Louis, School of Medicine, St Louis, Missouri
  - Palm Research Center, Las Vegas, Nevada
  - Columbia University Medical Center, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Allegheny Endocrinology Associates, Pittsburgh, Pennsylvania
  - Research Institute of Dallas, Dallas, Texas
- Germany (7):
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Frankfurt, Medizinische Klinik 1, Schwerpunkt Endokrinologie, Diabetologie, Ernährungsmedizin, Frankfurt
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Leipzig, Leipzig
  - LMU Clinic of University of Munich, Medical Clinic and Polyclinic IV, Munich
  - Medicover Neuroendokrinologie, Munich
  - Medicover Oldenburg MVZ, Oldenburg
- Greece (3):
  - General Hospital of Athens "Laiko", Endocrinology University Clinic, Athens
  - Aretaeio University Hospital Endocrinology Department, Faculty of Diabetes and Metabolism, Athens
  - General Hospital of Thessaloniki "Ippokratio", Thessaloniki
- Hungary (2):
  - Military Health Center, 2nd Department of Internal Medicine, Budapest
  - SZTE ÁOK I.sz. Belgyógyászati Klinika, Szeged
- Italy (5):
  - IRCCS Policlinico San Martino, Genova
  - Azienda Universitaria "Federico II", Napoli
  - Azienda Ospedaliera Padova, Department of Internal medicine, Padua
  - Policlinic Gemelli University Hospital IRCCS, Department of Endocrinology, Roma
  - AOUI Verona, Policlinic of GB Rossi, Verona
- Poland (4):
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Szpital Uniwersytecki w Krakowie, Krakow
  - Centrum Nowoczesnych Terapii "Dobry Lekarz", Krakow
  - Amicare Sp. z o.o. Sp. K., Lodz
  - Piekarskie Centrum Medyczne, Szpital Miejski, Piekary Śląskie
- Russia (7):
  - Interregional Clinical Diagnostic Center, Kazan'
  - "Atlas" Medical Center, Moscow
  - Sechenov Moscow First State Medical University, Moscow
  - Vladimirsky Moscow Regional Research Clinical Institute, Moscow
  - Novosibirsk State Regional Clinical Hospital, Novosibirsk
  - Interregional Clinical Diagnostic Center, Ryazan
  - Saratov Regional Clinic Hospital, Saratov
- Serbia (2):
  - Clinical Centre Serbia, Clinic for endocrinology, diabetes and metabolic diseases, Belgrade
  - Clinical Centre of Vojvodina, Clinic for endocrinology, diabetes and metabolic diseases, Novi Sad
- Spain (11):
  - University Hospital Complex A Coruña, A Coruña
  - University Hospital of Alicante, Alicante
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Clinic Barcelona, Barcelona
  - Hospital Universitario La Princesa, Madrid
  - Hospital Universitario Gregorio Marañón, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Complejo Hospitalario Universitario Santiago de Compostela, Santiago de Compostela
  - University Hospital Virgen del Rocio, Seville
  - Hospital Universitario y Politécnico La Fé, Valencia
  - Hospital Universitario de la Ribera, Valencia
- Turkey (Türkiye) (10):
  - Akdeniz University Faculty of Medicine Department of Endocrinology, Antalya
  - Aydın Adnan Menderes University Research and Application Hospital, Aydin
  - Pamukkale University Faculty of Medicine Department of Endocrinology, Denizli
  - Eskisehir Osmangazi University Medical Faculty, Eskişehir
  - Istanbul University Medical Faculty, Fatih
  - Kocaeli University Faculty of Medicine Department of Endocrinology and Metabolism, Kocaeli
  - Inonu University Medical Faculty Endocrinology Department, Malatya
  - Erciyes University Medical Faculty, Dept. of Endocrinology, Melikgazi
  - Karadeniz Technical University Farabi Hospital, Trabzon
  - Zonguldak Bulent Ecevit University Department of Internal Medicine, Division of Endocrinology and Metabolism Ibni Sina Campus, Zonguldak
- United Kingdom (5):
  - College of Medical and Dental Sciences, Birmingham
  - University Hospitals Coventry and Warwickshire NHS Trust, Coventry
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - The Christie NHS Foundation Trust, Manchester
  - Salford Royal Foundation Trust, Salford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Glatard A, Friberg-Hietala S, Keutzer L, Hansson A, Johnsson M, Tiberg F. Population Pharmacokinetic Analysis of an Octreotide Depot (CAM2029) in the Treatment of Acromegaly. Clin Pharmacokinet. 2025 Jul;64(7):1079-1092. doi: 10.1007/s40262-025-01522-3. Epub 2025 May 26. PMID 40418492